CLINICAL TRIAL: NCT00141648
Title: A Prospective Non-randomised Trial of Chemotherapy and Radiotherapy for Osteolymphoma
Brief Title: Chemotherapy and Radiotherapy for Osteolymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other); Australasian Radiation Oncology Lymphoma Group (Other); Wesley Research Institute (Other)
Responsible Party: Associate Professor David Christie, Trans Tasman Radiation Oncology Group (TROG)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 99.04; ALLG LY-02
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2009-10-01 (Estimated); Status verified 2009-09

CONDITIONS: Osteolymphoma
Keywords: Osteolymphoma; Chemotherapy; Radiotherapy; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; liposomal doxorubicin; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Chemotherapy followed by radiotherapy to begin 3 weeks after the last cycle.
  Interventions: Drug: Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone.; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cyclophosphamide, Doxorubicin, Vincristine, Prednisolone. — Given intravenously on days 1,11,43: Cyclophosphamide 750mg/m2, doxorubicin 50mg/m2, vincristine 1.4mg/m2. Given orally on days 1-5,22-27: Pednisolone 50mg/m2
  Other Names: Endoxan, Caelyx, Vincristine sulfate injection, Predsone
Radiation: Radiotherapy — Total 45 Gy in 25 fractions
  Other Names: Radiation

SUMMARY:
This trial is intended to determine the results obtained when standard treatment for Non Hodgkin's lymphoma is applied to the disease in a rare subtype which arises in bone. Patients in the study undergo a detailed assessment, then treatment with chemotherapy and radiotherapy, followed by close monitoring.

DETAILED DESCRIPTION:
Patients with non-Hodgkin's lymphoma arising primarily in bone have been studied using a number of different names making literature searching difficult. The term Osteolymphoma has been proposed to make searching easier in the future. Patients in this study undergoing staging which includes isotope bone scanning and PET scanning where available. Eligible patients then undergo treatment with three cycles of CHOP chemotherapy at conventional doses and shrinking field radiotherapy to a total of 45 Gy. Monoclonal antibodies are not included as good results have been obtained without using them. After treatment the patients are regularly monitored. The trial is presented twice per year at the meetings of TROG, ALLG and AROLG.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-Hodgkin's lymphoma in a bony site
* Limited extraosseous disease
* Ann Arbor stage IE
* Age >17
* ECOG performance status <3
* Expected survival > 6 months
* Patients capable of childbearing are using adequate contraception.
* Written informed consent

Exclusion Criteria:

* Previous radiotherapy
* Previous malignancy
* Medically unfit to undergo treatment

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2000-09; Primary Completion 2007-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Overall Survival. The time from registration to the date of death | Main analysis when accrual is complete at approx. 10 years.

SECONDARY OUTCOMES:
Time to local or regional failure. Measured from registration. | Main analysis when accrual is complete at approx. 10 years.
Pathological fracture rate. Measured from registration. | Main analysis when accrual is complete at approx. 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: David Christie, FRANZCR, Study Chair — East Coasr Cancer Centre
Locations (20):
- Australia (17):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - The Wesley Radiation Oncology Pty Ltd, Auchenflower, Queensland
  - Royal Brisbane Hospital, Herston, Queensland
  - Mater QRI, South Brisbane, Queensland
  - North Queensland Oncology Service, Townsville, Queensland
  - East Coast Cancer Centre, John Flynn Hospital, Tugun, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital, Launceston, Tasmania
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Andrew Love Cancer Care Centre, Geelong Hospital, Geelong, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Waikato Hospital, Hamilton
  - Palmerston North Hospital, Palmerston North

REFERENCES:
- [Background] Christie DR, Gabriel GS, Dear K. Adverse effects of a multicentre system for ethics approval on the progress of a prospective multicentre trial of cancer treatment: how many patients die waiting? Intern Med J. 2007 Oct;37(10):680-6. doi: 10.1111/j.1445-5994.2007.01451.x. PMID 17894765
- [Result] Christie D, Le T, Watling K, Cornes D, O'Brien P, Hitchins R. Quality assurance audit: a prospective non-randomised trial of chemotherapy and radiotherapy for osteolymphoma (TROG 99.04/ALLG LY02). J Med Imaging Radiat Oncol. 2009 Apr;53(2):203-6. doi: 10.1111/j.1754-9485.2009.02054.x. PMID 19527368
- [Derived] Christie D, Dear K, Le T, Barton M, Wirth A, Porter D, Roos D, Pratt G. Limited chemotherapy and shrinking field radiotherapy for Osteolymphoma (primary bone lymphoma): results from the trans-Tasman Radiation Oncology Group 99.04 and Australasian Leukaemia and Lymphoma Group LY02 prospective trial. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1164-70. doi: 10.1016/j.ijrobp.2010.03.036. Epub 2010 Jul 16. PMID 20638196
- See also: Click here for more information about this study on the TROG official website — http://www.trog.com.au